CLINICAL TRIAL: NCT02937077
Title: The Nordic Atrial Fibrillation and Stroke Study
Brief Title: Atrial Fibrillation in Cryptogenic Stroke and TIA
Acronym: NOR-FIB
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Ostfold Hospital Trust (Other); Haukeland University Hospital (Other); Rigshospitalet, Denmark (Other); Bispebjerg Hospital (Other); The Hospital of Vestfold (Other); Sykehuset Telemark (Other Government); Herlev Hospital (Other); Nordlandssykehuset HF (Other); Vestre Viken Hospital Trust (Other); Helse Stavanger HF (Other Government); Molde Hospital (Other); Drammen sykehus (Other); Diakonhjemmet Hospital (Other); University Hospital of North Norway (Other); Ullevaal University Hospital (Other); Sykehuset Innlandet HF (Other); Skane University Hospital (Other)
Responsible Party: Principal Investigator, Anne Hege Aamodt, Dr., Oslo University Hospital
Other Study IDs: 2013/2371
Record Dates: First submitted 2016-03-04; First posted 2016-10-18 (Estimated); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Atrial Fibrillation; Ischemic Stroke; TIA
Keywords: etiology
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Medtronic Reveal LINQ

SUMMARY:
Background:

Different studies with real-life data and randomized controlled trials have shown a detection rate of paroxysmal atrial fibrillation (AF) of 10-20% in patients with cryptogenic stroke using insertable continuous cardiac monitoring for 6 months. More studies are needed, however, to identify factors which can be used to select the patients where the possibility of detecting AF with prolonged rhythm monitoring is highest, to evaluate the best duration of rhythm monitoring, to determine the optimal deﬁnition of short-term AF that warrants intervention and to evaluate whether intervention results in improved clinical outcomes.

Methods: The NOR-FIB study is a multi-centre prospective observational trial, designed to evaluate detection of AF in cryptogenic stroke and transient ischemic attack (TIA). Patients admitted with cryptogenic stroke or TIA in stroke units in the Nordic countries, aged 18-80 years are included and have the Reveal LINQ® Insertable cardiac monitor system implanted for 12 months for the purpose of AF detection. Biomarkers that may identify patients, who could derive the most clinical benefit from the detection of AF by prolonged monitoring, are being studied.

Conclusion: This NOR-FIB study will increase our knowledge regarding the occurrence of AF in patients with cryptogenic stroke and TIA that potentially can improve secondary prevention. The study will provide information on biomarkers that may be used to select cryptogenic TIA and stroke patients for long-term monitoring as well as information on the significance of short-term AF and optimal duration of cardiac rhythm monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Cryptogenic ischemic stroke patients or symptomatic TIA < 21 days from symptom start.
2. A stroke/TIA is considered to be cryptogenic if no cause can be determined despite an extensive workup according to the standard protocol of the participating center. Before inclusion to the study, the following tests are required as standard tests to establish the diagnosis of cryptogenic stroke or TIA:

   1. Brain MRI or CT†
   2. 12-lead ECG for AF detection
   3. 24-h ECG monitoring for AF detection and premature atrial complex analysis (e.g. Holter)
   4. TEE (transesophageal echocardiography) highly recommended or TTE (transthoracic echocardiography)
   5. Colour Duplex ultrasound examination of the pre-cerebral arteries
   6. CTA or MRA of head and neck to rule out other causes of stroke pathologies
3. Age 18 to 80 at onset of TIA/stroke
4. A participation consent form signed by the patient or a legally authorized representative.

   * TIA cases with acute non-lacunar infarct on Diffusion Weighted Imaging are included as TIA events.

Exclusion Criteria:

1. Known etiology of TIA or stroke.
2. TIA without documented cerebral ischemia on Diffusion Weighed Imaging.
3. Untreated hyperthyroidism
4. Myocardial infarction less than 1 month prior to the stroke or TIA.
5. Coronary bypass grafting less than 1 month prior to the stroke or TIA.
6. Valvular heart disease requiring immediate surgical intervention.
7. History of atrial fibrillation or atrial flutter.
8. Patent Foramen Ovale (PFO) or PFO where there is or was an indication to start oral anticoagulation
9. Permanent indication for OAC treatment at enrollment.
10. Permanent contra-indication for OAC.
11. Life expectancy less than 1 year.
12. Pregnancy
13. An indication for an Implantable Pulse Generator (IPG), Implantable Cardioverter-Defibrillator (ICD), Cardiac Resynchronization Therapy (CRT) or an implantable hemodynamic monitoring system.
14. Patient otherwise not eligible for the study or adherent for follow-up (e.g. non-resident) or has concurrent disease which may affect clinical outcome (e.g. multiple sclerosis, cancer).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to stroke units with cryptogenic ischemic stroke or TIA
Sampling Method: Non-Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation detection rate | within 6 months

SECONDARY OUTCOMES:
AF detection rate | within 12 months
Levels of miRNAs related to atrial fibrillation | 12 months
Levels of NT-proBNP | baseline and 12 months
Levels of Troponin-T | baseline and 12 months
Levels of inflammation biomarkers | baseline and 12 months
Prestroke/pre-TIA CHA2DS2-VASc score | baseline
Incidence of recurrent stroke or TIA - percentage of stroke/TIA within 12 9. Incidence of recurrent stroke or TIA - percentage of stroke/TIA | 12 months
Use of oral anticoagulation - percentage of patients who are using OAC drugs | 12 months
Use of antiarrhythmic drugs - percentage of patients who are using antiarrhythmic drugs | 12 month
Health Outcome as Evaluated by an EQ-5D Questionnaire - EQ-5D quality of life score | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne Hege Aamodt, MD, PhD, Principal Investigator — Oslo University Hospital; Dan Atar, MD, PhD, Study Chair — Oslo University Hospital
Locations (2):
- Norway (2):
  - Østfold Hospital Trust, Sarpsborg, Grålum
  - Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: Yes
Plan to share IPD

REFERENCES:
- [Background] Li L, Yiin GS, Geraghty OC, Schulz UG, Kuker W, Mehta Z, Rothwell PM; Oxford Vascular Study. Incidence, outcome, risk factors, and long-term prognosis of cryptogenic transient ischaemic attack and ischaemic stroke: a population-based study. Lancet Neurol. 2015 Sep;14(9):903-913. doi: 10.1016/S1474-4422(15)00132-5. Epub 2015 Jul 27. PMID 26227434
- [Background] Tomson TT, Passman R. The Reveal LINQ insertable cardiac monitor. Expert Rev Med Devices. 2015 Jan;12(1):7-18. doi: 10.1586/17434440.2014.953059. Epub 2014 Aug 26. PMID 25154970
- [Background] Sanna T, Diener HC, Passman RS, Di Lazzaro V, Bernstein RA, Morillo CA, Rymer MM, Thijs V, Rogers T, Beckers F, Lindborg K, Brachmann J; CRYSTAL AF Investigators. Cryptogenic stroke and underlying atrial fibrillation. N Engl J Med. 2014 Jun 26;370(26):2478-86. doi: 10.1056/NEJMoa1313600. PMID 24963567
- [Background] Ziegler PD, Rogers JD, Ferreira SW, Nichols AJ, Sarkar S, Koehler JL, Warman EN, Richards M. Real-World Experience with Insertable Cardiac Monitors to Find Atrial Fibrillation in Cryptogenic Stroke. Cerebrovasc Dis. 2015;40(3-4):175-81. doi: 10.1159/000439063. Epub 2015 Aug 28. PMID 26314298
- [Background] Christensen LM, Krieger DW, Hojberg S, Pedersen OD, Karlsen FM, Jacobsen MD, Worck R, Nielsen H, Aegidius K, Jeppesen LL, Rosenbaum S, Marstrand J, Christensen H. Paroxysmal atrial fibrillation occurs often in cryptogenic ischaemic stroke. Final results from the SURPRISE study. Eur J Neurol. 2014 Jun;21(6):884-9. doi: 10.1111/ene.12400. Epub 2014 Mar 15. PMID 24628954
- [Background] Wu N, Chen X, Cai T, Wu L, Xiang Y, Zhang M, Li Y, Song Z, Zhong L. Association of inflammatory and hemostatic markers with stroke and thromboembolic events in atrial fibrillation: a systematic review and meta-analysis. Can J Cardiol. 2015 Mar;31(3):278-86. doi: 10.1016/j.cjca.2014.12.002. Epub 2014 Dec 9. PMID 25746020
- [Background] Howlett PJ, Hatch FS, Alexeenko V, Jabr RI, Leatham EW, Fry CH. Diagnosing Paroxysmal Atrial Fibrillation: Are Biomarkers the Solution to This Elusive Arrhythmia? Biomed Res Int. 2015;2015:910267. doi: 10.1155/2015/910267. Epub 2015 Jul 1. PMID 26229966
- [Derived] Ratajczak-Tretel B, Lambert AT, Al-Ani R, Arntzen K, Bakkejord GK, Bekkeseth HMO, Bjerkeli V, Eldoen G, Gulsvik AK, Halvorsen B, Hoie GA, Ihle-Hansen H, Ingebrigtsen S, Kremer C, Krogseth SB, Kruuse C, Kurz M, Nakstad I, Novotny V, Naess H, Qazi R, Rezaj MK, Rorholt DM, Steffensen LH, Somark J, Tobro H, Truelsen TC, Wassvik L, AEgidius KL, Atar D, Aamodt AH. Underlying causes of cryptogenic stroke and TIA in the nordic atrial fibrillation and stroke (NOR-FIB) study - the importance of comprehensive clinical evaluation. BMC Neurol. 2023 Mar 21;23(1):115. doi: 10.1186/s12883-023-03155-0. PMID 36944929